Alcon - Business Use Only Effective Date: 08-Mar-2019

Document: TDOC-0056081 Version: 1.0; CURRENT; Most-Recent; Effective

Status: Effective 

Title

# Clinical Comparison of DDT2 Contact Lens and a Daily Disposable Contact Lens - Study 2

Protocol Number: CLE383-C010/NCT03888482

Development Stage of

Sponsor Name and

Product Support

Project:

Alcon Research, Ltd. and its affiliates ("Alcon")

Address: 6201 South Freeway

Fort Worth, Texas 76134-2099

Test Product: DDT2 (Verofilcon A) contact lens

Property of Alcon Laboratories

Confidential

May not be used, divulged, published, or otherwise disclosed without the consent of

Alcon Laboratories


Status: Effective 

Effective Date: 08-Mar-2019

Investigator Agreement:

I have read the clinical study described herein, recognize its confidentiality, and
agree to conduct the described trial in compliance with Good Clinical Practice
(GCP), the ethical principles contained within the Declaration of Helsinki, this
protocol, all applicable regulatory authority regulations, and conditions of approval
imposed by the reviewing IRB or regulatory authority.

- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as
  described in the protocol, current Investigator's Brochure, product information, or
  other sources provided by the Sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements of the Sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| | Have you ever been disqualified as an Investigator by any Regulatory Authority? | | |
|---|---|---|---|
| | □ No □Yes | | |
| | Have you ever been | involved in a study or other research that was terminated | ? |
| | □ No □Yes | | |
| | If yes, please explain | n here: | |
| Pr | incipal Investigator: | | |
| | | Signature De | ate |
| | me and professional sition: | | |
| Ad | ldress: | | |
| | | Table of Contents | |
| Tab | le of Contents | | 2 |
| List | of Tables | | 5 |

| | | Siness Use Only OCC-0056081 Version: 1.0; CURRENT; Most-Recent; Effective Date: 08 | -Mar-2019 |
|---|---|---|---|
| | ocument: TD<br>atus: Effectiv | | age 3 of 55 |
| Li | st of Figur | res | 6 |
| 1 | GLOSS | ARY OF TERMS | 7 |
| 2 | LIST OF | F ACRONYMS AND ABBREVIATIONS | 12 |
| 3 | PROTO | COL SUMMARY | 14 |
| 4 | PROTO | COL AMENDMENTS | 22 |
| | 4.1 | Amendments | 22 |
| 5 | | DUCTION | |
| | 5.1 | Rationale and Background | 22 |
| | 5.2 | Purpose of the Study | |
| | 5.3 | Risks and Benefits | |
| 6 | STUDY | OBJECTIVES | 24 |
| | 6.1 | Primary Objective(s) | 24 |
| | 6.2 | Secondary Objective(s) | 24 |
| | 6.3 | | |
| | 6.4 | Safety Objective(s) | 24 |
| 7 | INVEST | TIGATIONAL PLAN | 25 |
| | 7.1 | Study Design | 25 |
| | 7.2 | Rationale for Study Design | 25 |
| | 7.3 | Rationale for Duration of Treatment/Follow-Up | 26 |
| | 7.4 | Rationale for Choice of Control Product | 26 |
| | 7.5 | Data Monitoring Committee | 26 |
| 8 | STUDY | POPULATION | 26 |
| | 8.1 | Inclusion Criteria | 26 |
| | 8.2 | Exclusion Criteria | 27 |
| | 8.3 | Rescreening of Subjects | 28 |
| 9 | TREATI | MENTS ADMINISTERED | 28 |
| | 9.1 | Investigational Product(s) | 28 |
| | 9.2 | Other Medical Device or Medication Specified for Use During the Stud | |
| | 9.3 | Treatment Assignment / Randomization | |
| | 9.4 | Treatment masking | 32 |

9.5

| A 1 | ъ. | TT. | $\sim$ 1 |
|-------|------------|-----|----------|
| Alcon | - Business | Use | Oniv |


Effective Date: 08-Mar-2019

| Sta | tus: Effective | ; | Page 4 | 01 55 |
|---|---|---|---|---|
| | 9.6 | Changes | to concomitant medications, treatments/ procedures | 35 |
| 10 | STUDY | PROCED | URES AND ASSESSMENTS | 35 |
| | 10.1 | Informed | l Consent and Screening | 35 |
| | 10.2 | Descripti | ion of Study Procedures and Assessments | 36 |
| | | 10.2.1 | Demographics | 36 |
| | | 10.2.2 | Medical History | 36 |
| | | 10.2.3 | Investigational Product Compliance | 36 |
| | | 10.2.4 | AE Collection: Safety Assessment | 36 |
| | | 10.2.5 | Slit-Lamp Biomicroscopy: Safety and Effectiveness Assessment | 36 |
| | | 10.2.6 | Device Deficiencies: Safety Assessment | |
| | 10.3 | Unsched | uled Visits | 37 |
| | 10.4 | Discontin | nued Subjects | 37 |
| | | 10.4.1 | Screen Failures | 37 |
| | | 10.4.2 | Discontinuations | |
| | | 10.4.3 | Schedule of Procedures and Assessments for Subjects Discontinue from Investigational Product | |
| | 10.5 | Clinical | Study Termination | |
| | | 10.5.1 | Follow-up of subjects after study participation has ended | |
| 11 | ADVERS | | TS AND DEVICE DEFICIENCIES | |
| | 11.1 | General 1 | Information | 39 |
| | 11.2 | Monitori | ng for Adverse Events | 40 |
| | 11.3 | Procedur | res for Recording and Reporting | 40 |
| | 11.4 | Return P | roduct Analysis | 43 |
| | | 11.4.1 | Alcon Marketed Product | 43 |
| | | 11.4.2 | Non-Alcon Marketed Product | 43 |
| | 11.5 | Unmaski | ing of the Study Treatment | 43 |
| | 11.6 | Follow-U | Jp of Subjects with Adverse Events | 43 |
| | 11.7 | Pregnand | ey in the Clinical Study | 44 |
| 12 | ANALYS | SIS PLAN | T | 44 |
| | 12.1 | Subject I | Evaluability | 44 |
| | 12.2 | Analysis | Sets | 45 |
| | | 12.2.1 | Safety Analysis Set | 45 |
| | | 12.2.2 | Full Analysis Set | 45 |
| | | 12.2.3 | Per Protocol Analysis Set | 45 |
| | 12.3 | Demogra | aphic and Baseline Characteristics | 45 |

| | | _ | _ | | | _ | | _ |
|--------|---|-----|-----|-----|-----|-------|-----|-----|
| Alcon | | Rп | cin | OCC | I C | a (1) | m | l 🔻 |
| AICUII | _ | Du. | эш | | | | 411 | ιv |

Effective Date: 08-Mar-2019

| Document: TDO<br>Status: Effective | | |
|---|---|---|
| 12.4 | Effectiveness Analyses | 45 |
| | 12.4.1 Analysis of Primary Effectiveness Endpoint(s) | 46 |
| | 12.4.1.1 Statistical Hypotheses | 46 |
| | 12.4.1.2 Analysis Methods | 46 |
| 12.5 | Handling of Missing Data | 48 |
| 12.6 | Safety Analyses | 49 |
| 12.7 | Interim Analyses and Reporting | 49 |
| 12.8 | Sample Size Justification | 50 |
| 13 DATA H | ANDLING AND ADMINISTRATIVE REQUIREMENTS | 50 |
| 13.1 | Subject Confidentiality | 50 |
| 13.2 | Completion of Source Documents and Case Report Forms | 51 |
| 13.3 | Data Review and Clarifications | 52 |
| 13.4 | Sponsor and Monitoring Responsibilities | 52 |
| 13.5 | Regulatory Documentation and Records Retention | 52 |
| 13.6 | Quality Assurance and Quality Control | 53 |
| 14 ETHICS | | 53 |
| 15 REFERE | ENCES | 55 |
| 15.1 | References applicable for all clinical studies | 55 |
| | 15.1.1 US references applicable for clinical studies | |
| 15.2 | References for this clinical study | 55 |
| | List of Tables | |
| Table 2–1 | List of Acronyms and Abbreviations Used in This Protocol | 12 |
| Table 3–1 | Schedule of Study Procedures and Assessments | 20 |
| Table 6–1 | Primary Objective(s) | 24 |
| Table 6–3 | Safety Objective(s) | 24 |
| Table 9–1 | Test Product | 28 |

| Alcon - Busi | Effective Date: 08-Mar-2019 | |
|---|---|---|
| Document: TDO Status: Effective | | |
| Table 9–2 | Control Product | 30 |
| Table 9–3 | Unmasked Individuals Associated with the Study | 32 |
| | List of Figures | |
| Figure 7–1 | Study Design | 25 |
| Figure 11–1 | Categorization of All AEs | 39 |
| Figure 11-2 | Categorization of All Serious AEs | 40 |


Status: Effective 

Effective Date: 08-Mar-2019

# 1 GLOSSARY OF TERMS

| Names of test product(s) | Throughout this document, test product(s) will be referred to as: DDT2 |
|---|---|
| Name of Control Product(s) | clariti® 1 day (Clariti 1 Day or Clariti) |
| Adverse Device Effect | Adverse event related to the use of an investigational |
| (ADE) | medical device (test product) or control product. Note: This |
| | definition includes adverse events resulting from insufficient |
| | or inadequate instructions for use, deployment, |
| | implantation, installation, or operation; any malfunction; |
| | and use error or intentional misuse of the test product or |
| | control product. |
| Adverse Event (AE) | Any untoward medical occurrence, unintended disease or |
| | injury, or untoward clinical signs (including abnormal |
| | laboratory findings) in subjects, users or other persons, |
| | whether or not related to the investigational medical device |
| | (test product). Note: For subjects, this definition includes |
| | events related to the test product, the control product, or the |
| | procedures involved. For users or other persons, this |
| | definition is restricted to events related to the test product. |
| | Requirements for reporting Adverse Events in the study can |
| | be found in Section 11. |
| Anticipated Serious | Serious adverse device effect, which by its nature, |
| Adverse Device Effect | incidence, severity, or outcome has been identified in the |
| | risk management file. |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, |
| | quality, durability, reliability, safety, or performance. Note: |
| | This definition includes malfunctions, use errors, and |
| | inadequate labeling. |
| | Requirements for reporting Device Deficiencies in the study can be found in Section 11. |

Version: 1.0; CURRENT; Most-Recent; Effective

Effective Date: 08-Mar-2019

Document: TDOC-0056081

Status: Effective 

| Enrolled Subject | Any subject who signs an informed consent form for participation in the study. |
|---|---|
| Interventional Clinical Trial | A research trial that prospectively assigns, whether |
| interventional emiliar Trial | randomly or not, human participants or groups of humans to one or more health-related interventions to evaluate the effects on health outcomes, and/or a research trial in which diagnostic or monitoring procedures beyond standard of care are conducted and generate outcomes for use in analysis of data. |
| Investigational Product | Is defined as a preventative (vaccine), a therapeutic (drug or biologic), device, diagnostic, or palliative used as a test or control product in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the authorized form, or when used for an unauthorized indication, or when used to gain further information about the authorized form. |
| Malfunction | Failure of a medical device to perform in accordance with its intended purpose when used in accordance with the instructions for use or clinical investigation plan. Performance specifications include all claims made in the labeling of the device. The intended performance of the device refers to the intended use for which the device is labeled or marketed. |
| Non-serious Adverse Event | Adverse event that does not meet the criteria for a serious adverse event. |
| Postmarketing/Post-<br>authorization study | Any study conducted within the conditions laid down in product labelling and other conditions laid down for the marketing of the product or under normal conditions of use. A postmarketing study falls either within the definitions of an interventional or a non-interventional study and may also fall within the definition of a post-approval study. |


Status: Effective 

Effective Date: 08-Mar-2019

| Product Complaints | Any oral, electronic, or written communication that alleges |
|---|---|
| | deficiencies related to the identity (labeling), quality, durability, reliability, safety, effectiveness, or performance of a marketed product, including failure of the product, labeling or packaging to meet specifications, whether or not the product is related to or caused the alleged deficiency. A complaint may allege that an adverse event or medical device malfunction has occurred. |
| Randomized Subjects | Any subject who is assigned a randomized treatment. |
| Serious Adverse Device | Adverse device effect that has resulted in any of the |
| Effect (SADE) | consequences characteristic of a serious adverse event. |
| Serious Adverse Event (SAE) | <ul> <li>Adverse event that led to any of the following:</li> <li>Death.</li> <li>A serious deterioration in the health of the subject that either resulted in: <ul> <li>a. a life-threatening illness or injury.</li> <li>Note: Life-threatening means that the individual was at immediate risk of death from the event as it occurred, ie, it does not include an event which hypothetically might have caused death had it occurred in a more severe form.</li> <li>b. any potentially sight-threatening event or</li> </ul> </li> </ul> |
| | b. any potentially sight-threatening event or permanent impairment to a body structure or a body function. |


Effective Date: 08-Mar-2019

Document: TDOC-0056081  Status: Effective

| Status: Effective | Fage 10 01 53 |
|---|---|
| | c. in-patient hospitalization or prolonged |
| | hospitalization. |
| | Note: Planned hospitalization for a pre- |
| | existing condition, without serious |
| | deterioration in health, is not considered a |
| | serious adverse event. In general, |
| | hospitalization signifies that the individual |
| | remained at the hospital or emergency ward |
| | for observation and/or treatment (usually |
| | involving an overnight stay) that would not |
| | have been appropriate in the physician's office |
| | or an out-patient setting. Complications that occur during hospitalization are adverse |
| | events. If a complication prolongs |
| | hospitalization or fulfills any other serious |
| | criteria, the event is serious. When in doubt as |
| | to whether "hospitalization" occurred, the |
| | event should be considered serious. |
| | <ul><li>d. a medical or surgical intervention to prevent</li><li>a) or b).</li></ul> |
| | <ul> <li>e. any indirect harm as a consequence of<br/>incorrect diagnostic test results when used<br/>within manufacturer's instructions for use.</li> </ul> |
| | • Fetal distress, fetal death, or a congenital abnormality |
| | or birth defect. |
| | Refer to Section 11 for additional SAEs. |
| | Refer to Section 11 for additional SALS. |
| Serious Public Health | Any event type which results in imminent risk of death, |
| Threat | serious deterioration in state of health, or serious illness that |
| | requires prompt remedial action. This would include: Events |
| | that are of significant and unexpected nature such that they |
| | become alarming as a potential public health hazard, eg, |
| | human immunodeficiency virus (HIV) or Bird Flu. |


Status: Effective 

Effective Date: 08-Mar-2019

| Significant Non-Serious Adverse Event | Is a symptomatic, device-related, non-sight threatening adverse event that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 11 for additional Significant Non-Serious AEs. |
|---|---|
| Unanticipated Serious<br>Adverse Device Effect | Serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the risk management file. |
| Use Error | Act or omission of an act that results in a different medical device response than intended by manufacturer or expected by user. Note: This definition includes slips, lapses, and mistakes. An unexpected physiological response of the subject does not in itself constitute a use error. |


Status: Effective 

Effective Date: 08-Mar-2019

# 2 LIST OF ACRONYMS AND ABBREVIATIONS

# Table 2-1 List of Acronyms and Abbreviations Used in This Protocol

| Abbreviation | Definition |
|---|---|
| ADE | Adverse device effect |
| AE | Adverse event |
| BCVA | Best corrected visual acuity |
| CFR | Code of Federal Regulations |
| CI | Confidence interval |
| Clariti 1 Day or | Clariti 1 Day Contact Lenses |
| Clariti | |
| COL | Clinical Operations Lead |
| CRF | Case report form |
| CSM | Clinical Site Manager |
| D | Diopter(s) |
| D/C | Discontinue |
| DDT2 | Daily Disposable T2 Contact Lenses |
| DEP | Deviations and evaluability plan |
| DT1 | DAILIES TOTAL1 Contact Lenses |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| EOD | End of day |
| FAS | Full analysis set |
| FDA | US Food and Drug Administration |
| GCP | Good Clinical Practice |
| GPCMS | Global Product Complaint Management System |
| HIV | Human immunodeficiency virus |
| IB | Investigator's Brochure |
| ICF | Informed consent form |
| ICH | International Council for Harmonization of Technical Requirements |
| | for Pharmaceuticals for Human Use |
| IEC | Independent ethics committee |
| IP | Investigational product |
| IRB | Institutional review board |
| IRT | Interactive response technology |
| ISO | International Organization for Standardization |
| logMAR | Logarithm of the minimum angle of resolution |
| LID | Lens identification |
| mm | Millimeter |
| MOP | Manual of procedures |
| n | Number |
| N/A | Not applicable |
| NI | Noninferiority |
| OD | Right eye |


Effective Date: 08-Mar-2019

Document: TDOC-0056081

 Status: Effective

| Abbreviation | Definition |
|--------------|-------------------------------|
| OS | Left eye |
| PP | Per protocol analysis set |
| SAE | Serious adverse event |
| SADE | Serious adverse device effect |
| SD | Standard deviation |
| SOP | Standard operating procedure |
| US | United States |
| VA | Visual acuity |


Effective Date: 08-Mar-2019

Document: TDOC-0056081  Status: Effective

# 3 PROTOCOL SUMMARY

| Investigational | Device |
|---|---|
| product type | |
| Study type | Interventional |
| Investigational | Test Product: DDT2 Contact Lens (Verofilcon A) (LID006841) |
| products | Control Product: Clariti 1 Day Contact Lens (somofilcon A) (LID014044) |
| | (LID014044) |
| Purpose and | The rationale for this study is to compare the objective and |
| rationale | subjective performance of DDT2 lenses to Clariti lenses. |
| Objective(s) | The primary objective of this study is to demonstrate |
| | noninferiority in the visual acuity (VA) at distance (distance VA) |
| | when wearing DDT2 contact lenses compared to Clariti contact |
| | lenses. |
| Endpoint(s) | Primary Effectiveness |
| | Distance VA (OD, OS; logMAR) |


Status: Effective 

Effective Date: 08-Mar-2019

| | Safety |
|---------------|------------------------------------------------------|
| | <ul><li>AEs</li><li>Biomicroscopy findings</li></ul> |
| | Device deficiencies |
| Assessment(s) | Effectiveness |
| | Distance VA (OD, OS; logMAR) |


Effective Date: 08-Mar-2019


Document: TDOC-0056081 Status: Effective


Status: Effective 

Effective Date: 08-Mar-2019

| Study Design Subject population | Safety • AEs • Biomicroscopy • Device deficiencies This is a prospective, randomized, crossover, double masked study comparing visual acuity with DDT2 contact lenses vs. Clariti contact lenses. Subjects will be expected to attend 3 study visits and wear study lenses for approximately 14 – 20 days (7 – 10 days for each study lens). Volunteer subjects aged 18 or over who are spherical soft contact lens wearers (excluding current/previous Clariti and DAILIES |
|---|---|
| | TOTAL1® (DT1) lens wearers), and for the last 3 months have |
| | worn their habitual lenses at least 5 days per week and at least 8 |
| | hours per day in daily wear modality. |
| | Planned number of subjects enrolled/consented: ~154 |
| | Planned number of completed subjects: 138 |
| Key inclusion | Current wearers of spherical soft contact lens who are 18 years of |
| criteria (See Section 8.1 for a | age or older. |
| complete list of | |
| inclusion criteria) | |
| Key exclusion | Previous or current habitual wearers of Clariti or DT1, or wear |
| criteria | habitual contact lenses in an extended wear fashion. |
| (See Section 8.2 for a | |
| complete list of | |
| exclusion criteria) | |

Version: 1.0; CURRENT; Most-Recent; Effective Document: TDOC-0056081

Status: Effective 

Effective Date: 08-Mar-2019

# Data analysis and **Planned Analysis** sample size To address the primary objectives, planned analyses are summarized below: justification Endpoint Comparison Statistical Method **Primary** Distance VA DDT2 vs Mixed effect repeated Clariti measures Noninferiority NI margin = 0.05 (logMAR)A sequential gatekeeping strategy followed by the Holm method will be implemented to control the testing of multiple effectiveness endpoints. No inferential testing will be performed for the effectiveness or safety analyses. **Sample Size Justification** Sample size calculations for distance VA endpoints, at 80% power, are summarized below: **Endpoint** Assumptions Type I error Primary Distance VA SD (paired difference) = 0.074One-sided 16 0.05 NI margin = 0.05

Document: TDOC-0056081


Effective Date: 08-Mar-2019

Status: Effective 

| Key words | Visual acuity, VA, daily disposable contact lenses |
|---|---|
| Associated materials | There are no associated materials with this study. Lubrication/rewetting drops will not be permitted. |

Alcon - Business Use Only Document: TDOC-0056081 Status: Effective

Table 3-1 **Schedule of Study Procedures and Assessments** 

| Procedure / Assessment | Visit 1 Screening / Baseline / Dispense Lens 1 (Lens 1 to be worn after washout period) | Visit 2<br>1-Week Follow-up<br>Lens 1 at EOD□ /<br>Dispense Lens 2 | Visit 3<br>1-Week Follow-up<br>Lens 2 at EOD□ / Exit | Unscheduled Visit /<br>Early Exit |
|---|---|---|---|---|
| | Washout period: Subjects will<br>discontinue habitual lens wear<br>after the screening visit until<br>the next day when they<br>commence wearing study<br>Lens 1∞ | 8 (-1/+2) days after Visit 1 Washout period: Subjects will wear spectacles after Visit 2 until the next day when they commence wearing study Lens 2.∞ | 8 (-1/+2) days after Visit 2 | N/A |
| Informed Consent | ✓ | - | - | - |
| Demographics | ✓ | - | - | - |
| Medical History | ✓ | ✓ | ✓ | ✓ |
| Concomitant Medications | ✓ | ✓ | ✓ | ✓ |
| Inclusion / Exclusion | ✓ | - | - | - |
| Habitual lens information (brand, power)* | ✓ | - | - | - |
| VA with habitual contact lens correction (OD, OS, Snellen distance)* | ✓ | - | ✓ (Exit procedure) | (✔) |
| BCVA (Snellen distance with manifest refraction) OD, OS* | <b>✓</b> | (✓) | (✓) | (*) |
| Biomicroscopy | ✓ | ✓ | ✓ | ✓ |
| Fit both study products (lenses) using fitting guide | ✓ | - | - | - |
| Dispense (provide) study lenses | ✓ | ✓ | - | (✔) |
| VA (logMAR distance) with study lenses, OD, OS | ✓* (with both fitting set lens types) | <b>√</b> | ✓ | (*) |

Print Date:

| Procedure / Assessment | Visit 1 Screening / Baseline / Dispense Lens 1 (Lens 1 to be worn after washout period) | Visit 2<br>1-Week Follow-up<br>Lens 1 at EOD□ /<br>Dispense Lens 2 | Visit 3<br>1-Week Follow-up<br>Lens 2 at EOD□ / Exit | Unscheduled Visit /<br>Early Exit |
|---|---|---|---|---|
| | Washout period: Subjects will<br>discontinue habitual lens wear<br>after the screening visit until<br>the next day when they<br>commence wearing study<br>Lens 1∞ | 8 (-1/+2) days after Visit 1 Washout period: Subjects will wear spectacles after Visit 2 until the next day when they commence wearing study Lens 2.∞ | 8 (-1/+2) days after Visit 2 | N/A |
| | • | | | • |
| | I | <b>–</b> | | I |
| AEs Device Deficiencies | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> |
| Exit Form | (✓) | (✓) | (✓) | (✓) |

<sup>□</sup> End of Day (8 – 16 hours of wear) \* source only (✓) assessment performed as necessary, eg, decrease of VA by 2 lines or more with investigational product (IP)

<sup>†</sup> Time points +/- 15 minutes


Status: Effective 

Effective Date: 08-Mar-2019

#### 4 PROTOCOL AMENDMENTS

Modification of the protocol is prohibited without prior written agreement in the form of a protocol amendment. All amendments must be created by the Study Sponsor and must be approved by the IRB/IEC and global and regional Health Authorities, as applicable, prior to implementation except when required to mitigate immediate safety risks or when the changes involve only logistical or administrative revisions.

Amendments may necessitate that the informed consent and other study-related material be revised. If the consent form is revised, all subjects currently enrolled in the study must sign the approved, revised informed consent (re-consent), as required by the IRB/IEC.

#### 4.1 Amendments

There are no amendments. This is the first version of the protocol.

### 5 INTRODUCTION

## 5.1 Rationale and Background

A recent paper has demonstrated that soft contact lenses continue to dominate contact lens prescribing and in the year 2018, soft contact lenses accounted for over 90% of lens fits. (Morgan 2019). Furthermore, it was reported that almost 32% of soft contact lenses were prescribed in a daily disposable modality. DDT2 is a new daily disposable silicone hydrogel contact lens with a material that combines high oxygen transmissibility with a low modulus of elasticity. The lens was recently approved by the FDA and will be marketed as Precision1™ (verofilcon A) Soft Contact Lenses.

The rationale for this study is the need to compare the objective and subjective performance of the new DDT2 lenses to an already marketed daily disposable contact lens (Clariti).

The primary endpoint for this study was selected to fulfill the primary objective. Procedures for measurement of these endpoints were selected based on common practice for these assessments. The design of this study is justified based upon previous preclinical and clinical testing, as described within the package insert. Clariti contact lenses were chosen as the control product because these lenses have the same wear modality.

# 5.2 Purpose of the Study

The primary objective of this study is to demonstrate noninferiority in distance VA when wearing DDT2 contact lenses compared to Clariti contact lenses.


Status: Effective 

Effective Date: 08-Mar-2019

At the end of the study a clinical study report will be prepared in accordance with applicable

At the end of the study, a clinical study report will be prepared in accordance with applicable regulatory requirements and standards.

The results from this study may be submitted as an abstract to be presented at conferences or as a manuscript to a journal if the data generated are of scientific interest.

## 5.3 Risks and Benefits

Contact lenses have several benefits in that they may offer improved peripheral vision and the added convenience of not wearing spectacles. Material properties and design characteristics of DDT2 contact lens are features consistent with successful contact lens wear. Based upon the pre-clinical and existing clinical data, DDT2 is known to be non-toxic and biocompatible for on-eye use.

Clariti lenses are intended and marketed for daily wear use under a daily disposable wear modality; further details on any known potential risks and benefits can be found in the package insert.

Neither the DDT2 nor the Clariti contact lenses are intended for use with a cleaning/disinfecting solution, and the biocompatibility with lens care solutions and any associated clinical effects are unknown.

A summary of the known potential risks and benefits associated with DDT2 can be found in the package insert. Risks are minimized by compliance with the eligibility criteria and study procedures, and through close supervision by a licensed clinician during exposure to the study lenses. The potential harms associated with on-eye exposure to the new lens materials include toxicity response, blurred vision, and ocular discomfort. In general, the risks associated with the wear of DDT2 are anticipated to be similar to other marketed daily disposable soft contact lenses.

There may also be unknown risks to use of DDT2 contact lenses. Any risk to subjects in this clinical study will be minimized by compliance with the eligibility criteria and study procedures, clinical oversight and monitoring.

The site personnel will educate subjects on proper hygiene and lens handling, and compliance with the use of contact lenses according to the protocol. Subjects should be instructed not to


Status: Effective 

Effective Date: 08-Mar-2019

wear contact lenses while sleeping or swimming. The site personnel will also advise the subjects to remove contact lenses and return for prompt follow-up of symptoms, such as ocular discomfort, foreign body sensation, excessive tearing, vision changes, or hyperemia.

Refer to the package insert for additional information.

## 6 STUDY OBJECTIVES

# 6.1 Primary Objective(s)

Table 6–1 Primary Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| The primary objective of this study is to demonstrate noninferiority in distance VA when wearing DDT2 contact lenses compared to Clariti contact lenses. | Distance VA (OD, OS; logMAR) |

# 6.2 Secondary Objective(s)

Not applicable.



# 6.4 Safety Objective(s)

Table 6–3 Safety Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| Describe the safety profile of the investigational products | <ul><li>AEs</li><li>Biomicroscopy findings</li><li>Device deficiencies</li></ul> |

Status: Effective 

#### 7 INVESTIGATIONAL PLAN

# 7.1 Study Design

This is a prospective, randomized, crossover, double masked study evaluating VA with DDT2 contact lenses vs. Clariti contact lenses.

Subjects will be expected to attend 3 study visits and wear study lenses for approximately 14-20 days (7 – 10 days for each study lens).

Figure 7–1 Study Design

Visit 1
Screening / Baseline /
Dispense Lens 1

Visit 2
Follow-up Lens 1,
1 Week, EOD Visit
Dispense Lens 2

Visit 3 Follow-up Lens 2, 1 Week EOD Visit / Exit

Effective Date: 08-Mar-2019

# 7.2 Rationale for Study Design

This study will be a prospective, randomized, crossover, Investigator and subject-masked trial and will include washout periods. The crossover study design will ensure that the same subject is exposed to both the test and control lens materials; therefore both objective and subjective responses will be obtained for both the lenses from the same subject. The study will include only those subjects who are successful wearers of spherical soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day. This will avoid confounding subjective and safety responses in non-adapted subjects. Moreover, the subjects will not be permitted to use artificial tears/rewetting drops during the course of the study as this may confound the primary effectiveness variable. The study will exclude any habitual wearers of Clariti or DT1 in order to reduce potential bias of wearers to their habitual contact lenses. This study will also exclude subjects who for the last 3 months have worn contact lenses in an extended wear modality. This study aims to compare the performance of two daily disposable contact lenses, therefore, subjects wearing lenses in an extended wear modality will be excluded as extended wear modality is known to impact the ocular physiology.

Status: Effective 

Effective Date: 08-Mar-2019

## 7.3 Rationale for Duration of Treatment/Follow-Up

Subjects will wear the lenses in a daily disposable wear modality for 8 -1/+2 days. The lenses will be provided by a qualified unmasked study staff member in such a manner that the subject and the Investigator remain masked to the lens type. As both the lenses are daily disposable lenses, they will be prescribed to be used in a daily disposable modality. The subjects will be asked to wear the lenses for at least 7 days, therefore, they are likely to have adapted to the lens material prior to collecting objective and subjective measurements.

#### 7.4 Rationale for Choice of Control Product

Both DDT2 and Clariti are soft contact lenses and are to be prescribed for single use, daily disposable wear. Clariti contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

## 7.5 Data Monitoring Committee

Not applicable.

#### 8 STUDY POPULATION

The study population consists of male and female subjects age 18 years or older who are wearers of soft daily contact lenses. Subjects who wear contact lenses in extended wear modality or are previous or current wearers of Clariti or DT1 contact lenses will be excluded. The study aims to enroll approximately 154 subjects at approximately 8 sites in the US with a target of 138 completed subjects. Site-specific targets may vary based upon individual site capabilities. Estimated time needed to recruit subjects for the study is approximately 6 weeks.

#### 8.1 Inclusion Criteria

Written informed consent must be obtained before any study specific assessment is performed. Upon signing informed consent, the subject will be considered as enrolled in the study.

Subjects eligible for inclusion in this study must fulfill **all** of the following criteria:

- 1. Subject must be at least 18 years of age.
- Subject must be able to understand and must sign an ICF that has been approved by an IRB.


Status: Effective 

Effective Date: 08-Mar-2019

3. Willing and able to attend all scheduled study visits as required per protocol.

- 4. Successful wear of spherical soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day.
- 5. Manifest cylinder of  $\leq 0.75$  D in each eye.
- 6. Best corrected VA of 20/25 or better in each eye.
- 7. Able to wear contact lenses within a range of sphere power from -1.00 to -6.00 D (0.25 D steps) and VA of 20/25 or better in each eye with fitting set lenses.

#### 8.2 Exclusion Criteria

Subjects fulfilling any of the following criteria are not eligible for participation in this study.

- Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the Investigator.
- 2. Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator.
- History of ocular or intraocular surgery, including refractive surgery and/or irregular cornea.
- 4. Biomicroscopy findings at baseline that are moderate (Grade 3) or higher and/or corneal vascularization that is mild (Grade 2) or higher.
- 5. Current or history of pathologically dry eye in either eye that, in the opinion of the Investigator, would preclude contact lens wear.
- 6. Current or history of herpetic keratitis in either eye.
- 7. Eye injury in either eye within 12 weeks immediately prior to enrollment for this trial.
- 8. Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.
- 9. Any use of topical ocular medications and artificial tear or rewetting drops that would require instillation during contact lens wear.


Status: Effective 

Effective Date: 08-Mar-2019

- 10. Previous or current habitual wearers of Clariti or DT1.
- 11. History of intolerance, hypersensitivity, or allergy to any component of the study products.
- 12. The Investigator, his/her staff, family members of the Investigator, family members of the Investigator's staff, or individuals living in the households of the aforementioned persons may not participate in the study.
- 13. Participation of the subject in a clinical trial within the previous 10 days or currently enrolled in any clinical trial.

Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation. Pregnancy should be included in the Medical History section of the eCRF when a pregnant woman enters the study or if a woman becomes pregnant during the study. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case-by-case basis.

## 8.3 Rescreening of Subjects

Rescreening of subjects is not allowed in this study.

#### 9 TREATMENTS ADMINISTERED

# 9.1 Investigational Product(s)

Test Product(s): DDT2 contact lenses

Control Product(s) (If applicable): Clariti 1 Day contact lenses

Table 9–1 Test Product

| Test Product | DDT2 contact lenses |
|---|---|
| Lens Identification<br>Number | LID006841 |
| Marketed Name | Precision1 contact lenses |
| Manufacturer | Alcon Laboratories, Inc.<br>6201 South Freeway<br>Fort Worth, Texas 76134-2099<br>USA |

Version: 1.0; CURRENT; Most-Recent; Effective Document: TDOC-0056081

 Status: Effective

Effective Date: 08-Mar-2019

| Indication for use and intended purpose in the current study | The intended use of this product is for vision correction. |
|---|---|
| Product description<br>and parameters<br>available for this<br>study | Material: verofilcon A • Water content: 51% • Power range: -1.00 to -6.00 D, 0.25 D steps • Base curve: 8.3 mm • Diameter: 14.2 mm |
| Formulation | Refer to the package insert |
| Usage | Wear: Daily Wear Bilateral Replacement period: |
| | <ul> <li>Daily Disposable</li> <li>Exposure:</li> <li>Approximately 10 hours per day (8 - 16 hours), every day, over the study treatment duration (8 days -1/+2)</li> </ul> |
| | Lens Care: N/A |
| Number/Amount of product to be provided to the subject | Lenses will be provided in packages of approximately 12 lenses per box per power, identified with the following: - a color coded label stating the protocol number - LID Number - power - an investigational use only statement - tracking number |
| Packaging description | Blister foil pack |
| Labeling description | Blister foil label includes at a minimum: - lens identifier - base curve - diameter - manufacturing protocol number - packing solution - power - lot number - expiration date - content statement - investigational device statement - Sponsor information |


Status: Effective 

Effective Date: 08-Mar-2019

| Storage conditions | Stored at room temperature |
|--------------------|--------------------------------------------------|
| Supply | Alcon will provide fitting set and study lenses. |

## Table 9–2 Control Product

| Control Product(s) | Clariti 1 Day |
|---|---|
| Manufacturer | CooperVision® |
| Lens Identification<br>Number | LID014044 |
| Indication for Use | The intended use of this product is for vision correction. |
| Product description<br>and parameters<br>available for this<br>study | Material: somofilcon A • Water content: 56% • Power range: -1.00 to -6.00 D, 0.25 D steps • Base curve: 8.6 mm • Diameter: 14.1 mm |
| Formulation | Refer to package insert |
| Usage | <ul> <li>Wear: <ul> <li>Daily Wear</li> <li>Bilateral</li> </ul> </li> <li>Replacement period: <ul> <li>Daily Disposable</li> </ul> </li> <li>Exposure: <ul> <li>Approximately 10 hours per day (8 - 16 hours), every day, over the study treatment duration (8 days -1/+2)</li> </ul> </li> <li>Lens Care: N/A</li> </ul> |
| Number/Amount of Product to be Provided to the subject Packaging | Lenses will be provided in packages of approximately 12 lenses per box per power, identified with the following: - a color coded label stating the protocol number - LID Number - power - an investigational use only statement - tracking number Blister foil pack |
| description | |


Status: Effective 

Effective Date: 08-Mar-2019

| Labeling description | Blister foil labels include at a minimum: |
|---|---|
| | - lens identifier |
| | - power |
| | - base curve |
| | - diameter |
| | - lot number |
| | - packing solution |
| | - expiration date |
| | <ul> <li>content statement</li> </ul> |
| | <ul> <li>investigational use statement</li> </ul> |
| | <ul> <li>Sponsor information</li> </ul> |
| Storage conditions | Stored at room temperature |
| Supply | Alcon will provide fitting set and study lenses. |

More information on both lenses can be found in their respective package inserts.

# 9.2 Other Medical Device or Medication Specified for Use During the Study

No other medical devices or medications are required to be used in conjunction with the treatments during the clinical study.

## 9.3 Treatment Assignment / Randomization

Subjects will be randomized in a 1:1 ratio to receive treatment in a crossover sequence of DDT2 then Clariti or Clariti then DDT2, respectively.

Only after signing the ICF, a subject will be assigned a subject number by the electronic data capture system.

A randomization list will be generated using a validated system that automates the random assignment of treatment sequences to randomization numbers in the specified ratio. Subjects will be assigned treatment sequences according to the randomization list uploaded in the IRT system. The randomization list will be generated and maintained by the Study Sponsor.

At Visit 1, all eligible subjects will be randomized via the EDC/IRT integration system to one of the treatment sequences. The Investigator or delegate will access the respective system after confirming that the subject meets all the eligibility criteria. A randomization number will be automatically assigned to the subject according to the subject randomization list but


Status: Effective 

Effective Date: 08-Mar-2019

will not be communicated to the site user. The EDC/IRT integration system will inform the site user of the treatment sequence assignment to be dispensed to the subject.

## 9.4 Treatment masking

This study is double-masked, with subjects randomized to use DDT2 and Clariti in the assigned sequence for the duration of 2 weeks (1 week for each period). Subjects, the Investigator, and masked study personnel (site and Sponsor) will be masked to the assigned treatment sequence.

Table 9-3 Unmasked Individuals Associated with the Study

| Unmasked Individual | Extent of Unmasking | Rationale |
|---|---|---|
| Unmasked Study | The Unmasked Study | The Unmasked Study |
| Coordinator | Coordinator(s) will manage | Coordinator(s) will be |
| | IP inventory, as well as IP | unmasked to allow for |
| | administration. This | storage and dispensing, as |
| | individual will have access | well as accountability for all |
| | to IP supply, accountability | IP. |
| | logs, and other documents or | |
| | supplies pertaining to IP. | |
| | The unmasked coordinator | |
| | will also assist with device | |
| | deficiency and AE | |
| | reporting. | |
| Clinical Operations Lead | The COL will have access to | The COL will be unmasked |
| (COL) | IP supply, accountability | to allow for oversight of the |
| () | logs, and other documents or | CSM, in conjunction with |
| | supplies pertaining to IP. | all IP accountability tasks. |
| | This individual assist with | |
| | masked and unmasked data | |
| | reviews. | |
| Clinical Site Manager | CSM will have access to IP | The CSM will be unmasked |
| (CSM) | supply, accountability logs, | to allow for performance of |
| | and other documents or | IP accountability, |
| | supplies pertaining to IP | management of device |
| | accountability. This | deficiencies and related AE |


Status: Effective 

Effective Date: 08-Mar-2019

| Unmasked Individual | Extent of Unmasking | Rationale |
|---|---|---|
| | individual monitors<br>unmasked and masked study<br>data. | lens returns, and other IP related tasks. |
| Clinical Supplies Coordinator | The Clinical Supplies Coordinator will have access to the IP inventory, accountability logs and other documents or supplies for management and reconciliation of the IP. | The Clinical Supplies Coordinator will be unmasked to allow for storage, management, and distribution of IP inventory and other IP related products/tasks. |
| Unmasked Data Manager(s) | The Unmasked Data Manager(s) will have access to restricted fields in EDC that would contain unmasking data. | The Unmasked Data Manager(s) will be unmasked to allow for review of all restricted data. |
| IRT Manager | The IRT Manager will be unmasked to allow for system programming, testing, and to allow for technical oversight of the system. | The IRT manager is unmasked to all aspects of the trial for system development purposes. |
| Randomization Specialist | The Randomization Specialist will be unmasked to allow for generation of the randomization list and uploading of that list into the IRT system. | Generates and therefore has full knowledge of treatment codes but otherwise is operationally not associated with the Clinical Trial Team or any decision-making aspects related to clinical trial design, execution, or reporting. |


Status: Effective 

Effective Date: 08-Mar-2019

This level of masking will be maintained throughout the conduct of the study. Unmasking will occur only after all planned study data have been validated, and the database locked.

Masked study personnel must avoid seeking information that may compromise masking. Unmasked study personnel must not disseminate information that is potentially unmasking to any masked personnel. The masked and unmasked site personnel must coordinate all study activities as necessary to protect masking and minimize bias during the study.

In the event of a medical emergency where the knowledge of subject treatment is required, an individual Investigator will have the ability to unmask the treatment assignment for a specific subject after contacting an appropriate Study Sponsor representative if time allows.

Unmasking must be done according to the instructions provided for the study IRT system.

Refer to Section 11.5.

## 9.5 Accountability Procedures

Upon receipt of the IPs, the Investigator or delegate must conduct an inventory. During the study, the masked Investigator must designate unmasked staff to provide the IPs to the subjects in accordance with their randomization assignment. Throughout the study, the Investigator or delegate must maintain records of IP dispensation and collection for each subject. This record must be made available to the study monitor for the purposes of verifying the accounting of IP supplies. Any discrepancies and/or deficiencies between the observed disposition and the written account must be recorded along with an explanation. All IPs sent to the Investigator must be accounted for by Study Sponsor personnel, and in no case be used in an unauthorized situation.

It is the Investigator's responsibility to ensure that:

- All study products are accounted for and not used in any unauthorized manner
- All used foils and unused supplies are returned by each subject
- All unused products are available for return to the Study Sponsor, as directed
- Any study lenses associated with a device deficiency or with any product-related AE
  (ie, ADE or SADE) are returned to the Study Sponsor for investigation, unless
  otherwise directed by the Sponsor. Refer to Section 11 of this protocol for additional
  information on the reporting of device deficiencies and AEs and the return of study
  products associated with these events.

The Investigator is responsible for proper disposition of all unused IPs at the conclusion of the study, according to the instructions provided in the MOP.


Effective Date: 08-Mar-2019

Document: TDOC-0056081

Status: Effective 

#### 9.6 Changes to concomitant medications, treatments/procedures

After the subject is enrolled into the study, the Investigator must instruct the subject to notify the study site about:

- Any new medications
- Alterations in dose or dose schedules for current medications
- Any medical procedure or hospitalization that occurred or is planned
- Any non-drug therapies (including physical therapy and blood transfusions)

The Investigator must document this information in the subject's case history source documents.

#### 10 STUDY PROCEDURES AND ASSESSMENTS

Subjects will be expected to attend 3 office visits over a period of approximately 2 weeks. Study lenses will be provided to the subjects to take home for daily wear during the course of the trial.

Study randomization will occur at Visit 1 with assigned lenses provided to take home at Visit 1 and Visit 2. Study contact lens fitting will occur at Visit 1 for both study lenses. If a subject cannot be successfully fit (either study lens) according to the study lens fitting guides as determined by the Investigator, they will be considered a screen failure and exited from the study.

will be conducted as outlined in the MOP. Worn Study tests, procedures, study contact lenses will be disposed of by the subject and used lidding foils will be returned to the site.

## 10.1 Informed Consent and Screening

The Investigator or delegate must explain the purpose and nature of the study, and have the subject read, sign, and date the IRB/IEC-approved informed consent document. The subject must sign the ICF BEFORE any study-specific procedures or assessments can be performed, including study-specific screening procedures. Additionally, have the individual obtaining consent from the subject and a witness, if applicable, sign and date the informed consent document.


Status: Effective 

Effective Date: 08-Mar-2019

The Investigator or delegate must provide a copy of the signed document to the subject and place the original signed document in the subject's chart, or provide documentation as required by local regulations.

## 10.2 Description of Study Procedures and Assessments

Detailed descriptions of assessments and procedures are provided in the MOP. The Investigator is responsible for ensuring responsibilities for all procedures and assessments are delegated to appropriately qualified site personnel.

## 10.2.1 Demographics

Obtain demographic information including age, race, ethnicity, and sex.

## **10.2.2 Medical History**

Collect medical history information, including information on all medications used within the past 30 days. Include herbal therapies, vitamins, and all over-the-counter as well as prescription medications. Throughout the subject's participation, obtain information on any changes in medical health and/or the use of concomitant medications.

## 10.2.3 Investigational Product Compliance

Review subject compliance with the IP usage and collect all used lidding foils, unused study IPs, and other products that were dispensed.

# 10.2.4 AE Collection: Safety Assessment

Assess and record any AEs that are observed or reported, including those associated with changes in concomitant medication dosing since the previous visit.

# 10.2.5 Slit-Lamp Biomicroscopy: Safety and Effectiveness Assessment

A slit-lamp exam must be performed on both eyes at every visit.

# 10.2.6 Device Deficiencies: Safety Assessment

Assess and record any device deficiencies that are reported or observed, including those associated with changes in concomitant medication dosing since the previous visit. Requirements for reporting device deficiencies in the study can be found in Section 11. Device deficiencies on comparator lenses should be reported per their manufacturer's guidelines.

Status: Effective 

Effective Date: 08-Mar-2019

#### 10.3 Unscheduled Visits

If a subject visit occurs between any regularly scheduled visits, this visit must be documented as an Unscheduled Visit. During all unscheduled visits, the Investigator must conduct the following procedures:

- Collect AE and device deficiency information
- Assess and record changes in medical condition or concomitant medication
- Perform biomicroscopy (assessments with or without study lenses, as applicable)
- Assess and record VAs, as necessary
- Perform lens surface and fitting assessments (study lenses) as applicable

The Investigator may perform additional procedures for proper diagnosis and treatment of the subject. The Investigator must document this information in the subject's case history source documents.

If during an Unscheduled Visit the subject is discontinuing the IP or discontinuing from the study, the Investigator must conduct Exit procedures according to Table 3-1 Schedule of Study Procedures and Assessments, as possible.

# 10.4 Discontinued Subjects

#### 10.4.1 Screen Failures

Screen failures are subjects who are excluded from the study after signing the informed consent and prior to randomization. This includes subjects who are unable to be fit for study lenses using the fitting guide.

The Investigator must document the reason for screen failure in the subject's case history source documents.

Subject numbers must not be re-used.

#### 10.4.2 Discontinuations

Discontinued subjects are individuals who voluntarily withdraw or are withdrawn from the study by the Investigator after signing informed consent, including screen failures.

Subject numbers of discontinued subjects must not be re-used.


Status: Effective 

Effective Date: 08-Mar-2019

Subjects may discontinue from the study or study treatment at any time for any reason. Subjects may also be discontinued from study treatment at any time if, in the opinion of the Investigator, continued treatment poses a risk to their health.

For subjects discontinuing from the study, the Investigator must complete all Exit procedures according to Table 3-1, Schedule of Study Procedures and Assessments, if the subject is willing and able, and if in the opinion of the Investigator it is safe for the subject to do so.

The Investigator must document the reason for study or treatment discontinuation in the subject's case history source documents.

To ensure the safety of all subjects who discontinue early, Investigators must assess each subject and, if necessary, advise them of any therapies and/or medical procedures that may be needed to maintain their health.

# 10.4.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product

Any subject discontinued from IP will be discontinued from the study and follow exit procedures.

# 10.5 Clinical Study Termination

The Study Sponsor reserves the right to close the investigational site or terminate the study in its entirety at any time.

If the clinical study is prematurely terminated or suspended by the Study Sponsor:

- The Study Sponsor must:
  - Immediately notify the Investigator(s) and subsequently provide instructions for study termination.
  - Inform the Investigator and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension.
- The Investigator must:
  - Promptly notify the IRB/IEC of the termination or suspension and of the reasons.
  - Provide subjects with recommendations for post-study treatment options as needed.

Effective Date: 08-Mar-2019

Document: TDOC-0056081

Status: Effective 

The Investigator may terminate the site's participation in the study for reasonable cause.

# 10.5.1 Follow-up of subjects after study participation has ended

Following this study, the subject will return to their eye care professional for their routine eye care.

#### 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### 11.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test article). Refer to the Glossary of Terms and figures below for categories of AEs and SAEs.

Figure 11-1 Categorization of All AEs



Status: Effective 

Effective Date: 08-Mar-2019

Figure 11-2 Categorization of All Serious AEs



#### **Device Deficiencies**

A device deficiency may or may not be associated with subject harm (ie, ADE or SADE); however, not all ADEs or SADEs are due to a device deficiency. The Investigator should determine the applicable category for the identified or suspect device deficiency and report any subject harm separately.

# 11.2 Monitoring for Adverse Events

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the Investigator should inquire about AEs by asking the standard questions:

- "Have you had any health problems since your last study visit?"
- "Have there been any changes in the medicines you take since your last study visit?"

Changes in *any protocol-specific parameters* evaluated during the study are to be reviewed by the Investigator. Any untoward (unfavorable and unintended) change in *a protocol-specific parameter* that is clinically relevant, in the opinion of the Investigator, is to be reported as an AE. These clinically relevant changes will be reported regardless of causality.

# 11.3 Procedures for Recording and Reporting

AEs are collected from the time of informed consent Any pre-existing medical conditions or signs/symptoms present in a subject prior to the start of the study (ie, before informed


Status: Effective 

Effective Date: 08-Mar-2019

consent is signed) are not considered AEs in the study and should be recorded in the Medical History section of the eCRF.

In addition, temporary lens awareness or visual changes during the fitting process are not considered AEs if the Investigator assesses that the symptom(s) can reasonably resolve within the anticipated adaptation period.

For each recorded event, the ADEs and SAEs documentation must include: date of occurrence, severity, treatment (if applicable), outcome, and assessments of the seriousness and causality. In addition, the Investigator must document all device deficiencies reported or observed with test and control articles on the Device Deficiency eCRF. The site must submit all available information on ADEs, SAEs, and device deficiencies to the Study Sponsor immediately as follows:

- ADEs or SAEs are documented on the Serious Adverse Event and Adverse Device Effect eCRF within 24 hours of the Investigator's or site's awareness.
- Device deficiencies are documented on the Device Deficiency eCRF within 24 hours of the Investigator's or site's awareness.
- A printed copy of the completed Serious Adverse Event and Adverse Device Effect and/or Device Deficiency eCRF must be included with product returns. Refer to the MOP for additional information on product returns.
- Additional relevant information after initial reporting must be entered into the eCRF as soon as the data become available.
- Document any changes to concomitant medications on the appropriate eCRFs.
- Document all relevant information from Discharge Summary, Autopsy Report,
   Certificate of Death, etc, if applicable, in narrative section of the Serious Adverse
   Event and Adverse Device Effect eCRF.

Note: Should the EDC system become non-operational, the site must complete the appropriate paper Serious Adverse Event and Adverse Device Effect and/or Device Deficiency Form. The completed form is faxed or emailed to the Study Sponsor at 1-817-302-1927 or MSUS.safety@alcon.com according to the timelines outlined above; however, the reported information must be entered into the EDC system once it becomes operational.


Status: Effective 

Effective Date: 08-Mar-2019

Study Sponsor representatives may be contacted for any protocol related question and their contact information is provided in the Manual of Procedures that accompanies this protocol (page 1).

Further, depending upon the nature of the AE or device deficiency being reported, the Study Sponsor may request copies of applicable portions of the subject's medical records. The Investigator must also report all AEs and device deficiencies that could have led to a SADE according to the requirements of regulatory authorities or IRB/IEC.

## **Intensity and Causality Assessments**

Where appropriate, the Investigator must assess the intensity (severity) of the AE based on medical judgment with consideration of any subjective symptom(s), as defined below:

#### Intensity (Severity)

Mild An AE is mild if the subject is aware of but can easily tolerate the sign or

symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort significant

enough to cause interference with the subject's usual activities.

Severe An AE is severe if the sign or symptom is incapacitating and results in the

subject's inability to work or engage in their usual activities.

For every AE in the study, the Investigator must assess the causality (Related or Not Related to the medical device or study procedure). An assessment of causality will also be performed by Study Sponsor utilizing the same definitions, as shown below:

#### Causality

Related An AE classified as related may be either definitely related or possibly related

where a direct cause and effect relationship with the medical device or study procedure has not been demonstrated, but there is a reasonable possibility that

the AE was caused by the medical device or study procedure.

Not Related An AE classified as not related may either be definitely unrelated or simply

unlikely to be related (ie, there are other more likely causes for the AE).


Status: Effective 

Effective Date: 08-Mar-2019

The Study Sponsor will assess the AEs and may upgrade the Investigator's assessment of seriousness and/or causality. The Study Sponsor will notify the Investigator of any AEs that is upgraded from non-serious to serious or from unrelated to related.

# 11.4 Return Product Analysis

Study Sponsor representatives and their contact information are provided in the MOP that accompanies this protocol.

#### 11.4.1 Alcon Marketed Product

Alcon products associated with device deficiencies and/or product related AEs should be returned and must include the Complaint # which will be provided by Study Sponsor after the case is entered in the Study Sponsor's Global Product Complaint Management System (GPCMS).

#### 11.4.2 Non-Alcon Marketed Product

When study products include non-Alcon marketed products, and such products are associated with device deficiencies and/or product related AEs, in the Investigator should report complaints directly to the manufacturer as per the manufacturer's instructions or local regulatory requirements, if applicable.

# 11.5 Unmasking of the Study Treatment

Masked information on the identity of the assigned medical device should not be disclosed during the study (see Section 9.4). If the treatment code needs to be broken in the interest of subject safety, the Investigator is encouraged to contact an appropriate Study Sponsor representative prior to unmasking the information if there is sufficient time. Dependent upon the individual circumstances (ie, medical emergency), the code may be broken prior to contact with the Study Sponsor. The Study Sponsor must be informed of all cases in which the code was broken and of the circumstances involved. Additionally, the Study Sponsor may be required to unmask the information in order to fulfill expedited regulatory reporting requirements.

# 11.6 Follow-Up of Subjects with Adverse Events

The Investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study.


Status: Effective 

Effective Date: 08-Mar-2019

The Investigator should provide the Study Sponsor with any new safety information (which includes new AEs and changes to previously reported AEs) that may affect the safety evaluation of the device. For AEs that are unresolved/ongoing at time of subject exit from study, any additional information received at follow-up should be documented in the eCRFs up to study completion (ie, database lock).

Any additional data received up to 1 month after subject discontinuation or exit must be documented and available upon the Study Sponsor's request. All complaints received after this time period will be considered and processed as spontaneous (following the postmarket vigilance procedures) and should be communicated to the medical device's manufacturer as per local requirements.

The Investigator should also report complaints on non-Alcon products directly to the manufacturer as per the manufacturer's instructions or local regulatory requirements.

# 11.7 Pregnancy in the Clinical Study

Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation. Pregnancy should be included in the Medical History section of the eCRF when a pregnant woman enters the study or if a woman becomes pregnant during the study. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case-by-case basis.

#### 12 ANALYSIS PLAN

Continuous variables will be summarized using the number of observations, mean, standard deviation (SD), median, minimum, and maximum, as well as confidence intervals (CIs) or confidence limits where applicable. Categorical variables will be summarized with counts and percentages from each category. Any deviations to the analysis plan will be updated during the course of the study as part of a protocol amendment or will be detailed in the clinical study report.

# 12.1 Subject Evaluability

Final subject evaluability must be determined prior to breaking the code for masked treatment sequence assignment and locking the database, based upon the Deviations and Evaluability Plan (DEP).


Status: Effective 

Effective Date: 08-Mar-2019

## 12.2 Analysis Sets

## 12.2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study, except for the lenses used at Visit 1 for the purpose of parameter optimization and fitting, as they are not intended for the assessment of safety. For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed in the corresponding lens sequence.

#### 12.2.2 Full Analysis Set

The full analysis set (FAS) is the set of all randomized subjects who are exposed to any study lenses evaluated in this study, except for the lenses used for optimization and fitting.

#### 12.2.3 Per Protocol Analysis Set

The per protocol (PP) analysis set is a subset of FAS and excludes all data/subjects that have met any of the critical deviation or evaluability criteria identified in the DEP. **Demographic** and Baseline Characteristics

Demographic and baseline characteristics will be summarized by lens sequence and overall. Counts and percentages will be presented for categorical variables such as sex, age group, race, and ethnicity. Number of observations, mean, SD, median, minimum, and maximum will be presented for continuous variables such as age.

# 12.4 Effectiveness Analyses

| This study defines 1 primary, |
|---|
| endpoint. All effectiveness evaluations will use the FAS as the primary analysis set. |
| The primary endpoint of distance VA will be tested at one-sided $\alpha$ =0.05 for noninferiority |

Print Date:


Status: Effective 

Effective Date: 08-Mar-2019

## 12.4.1 Analysis of Primary Effectiveness Endpoint(s)

The primary objective of this study is to demonstrate noninferiority in distance VA when wearing DDT2 contact lenses compared to Clariti contact lenses. The primary endpoint is distance VA with study lenses, collected for each eye in logMAR

# 12.4.1.1 Statistical Hypotheses

The null and alternative hypotheses are formulated in terms of the predefined margin of 0.05 for noninferiority:

$$H_0$$
:  $\mu_{(T)} - \mu_{(C)} \ge 0.05$   
 $H_a$ :  $\mu_{(T)} - \mu_{(C)} < 0.05$ 

where  $\mu_{(T)}$  and  $\mu_{(C)}$  denote the mean distance VA for DDT2 and Clariti, respectively, on the logMAR scale.

# 12.4.1.2 Analysis Methods

A mixed effect repeated measures model will be utilized to test these hypotheses. The model will include terms for lens, visit, lens by visit interaction, period, and sequence. Withinsubject correlation due to eye and the crossover design will also be accounted for in the model. Lens difference (DDT2 minus Clariti) and the corresponding one-sided 95% upper confidence limit will be computed. Noninferiority in distance VA will be declared if upper confidence limit is less than 0.05.



Version: 1.0; CURRENT; Most-Recent; Effective Document: TDOC-0056081

Effective Date: 08-Mar-2019


Status: Effective

Status: Effective


Effective Date: 08-Mar-2019


# 12.5 Handling of Missing Data

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out for the primary analyses.


Status: Effective 

Effective Date: 08-Mar-2019

# 12.6 Safety Analyses

The safety endpoints are:

- AEs
- Biomicroscopy findings
- Device deficiencies

There are no safety hypotheses planned in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of adverse events as well as the other listed parameters.

All AEs occurring from the time a subject signs informed consent to study exit will be accounted for in the reporting. Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. Descriptive summaries (counts and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities Preferred Terms. AEs leading to study discontinuation, significant non-serious AEs, and SAEs will be identified. Individual subject listings will be provided, as necessary.

Individual subject listings will be provided for AEs that occur after signing informed consent but prior to exposure to IP.

Each biomicroscopy parameter will be tabulated by its grade. For each biomicroscopy parameter, counts and percentages of eyes that experience an increase of  $\geq 2$  grades from baseline (last assessment prior to study lens exposure) to any subsequent visit within the same period will be presented. A supportive listing will be generated which will include all biomicroscopy data from all visits within the same period for those eyes experiencing the increase.

Two listings for device deficiencies, prior to exposure of study contact lenses and treatmentemergent, will be provided. Additionally, each device deficiency category will be tabulated.

No inferential testing will be done for safety analysis.

# 12.7 Interim Analyses and Reporting

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination.


Effective Date: 08-Mar-2019

Document: TDOC-0056081

Status: Effective 

## 12.8 Sample Size Justification

Sample size calculation is based on a prior clinical study (CLE383-C006) which evaluated performance of DDT2 and Clariti.

#### Primary Effectiveness

To demonstrate noninferiority (margin = 0.05 in logMAR; ½ line in Snellen) in distance VA as a one-tailed hypothesis with  $\alpha$ =0.05, and using a standard deviation of 0.074 for paired differences, 80% power can be attained with a sample size of 16 (8 per sequence).



# 13 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS

# 13.1 Subject Confidentiality

The Investigator must ensure that the subject's anonymity is maintained throughout the course of the study. In particular, the Investigator must keep an enrollment log with confidential identifying information that corresponds to the subject numbers and initials of each study participant. At the end of the clinical study, the Study Sponsor will collect a copy of the enrollment log without any identifying subject information. All documents submitted to the Study Sponsor will identify the subjects exclusively by number and demographic information. No other personally identifying information will be transmitted to the Study Sponsor.

The Study Sponsor may release anonymized study data to external researchers for purposes of future research directly related to the study objectives, or future research that is beyond the


Status: Effective 

Effective Date: 08-Mar-2019

scope of the current study objectives. The Informed Consent Form explains this to study subjects. Anonymization means that all identifiable information will be removed from the dataset and all links to the subjects in the study will be removed. Anonymization of the data will maintain confidentiality of the subjects who participate in the study so that they cannot be identified by external researchers. The anonymized data set will contain records from all of the subjects in the current study, but the anonymization process might change the data set in some ways, so external researchers will be informed that they might not be able to duplicate some of the results from this study.

## 13.2 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the CRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Site monitors are appointed by the Study Sponsor and are independent of study site staff.

If electronic records are maintained, the method of verification must be determined in advance of starting the study.

At a minimum, source documents include the following information for each subject:

- Subject identification (name, sex, race/ethnicity)
- Documentation of subject eligibility
- Date of informed consent
- Dates of visits
- Documentation that protocol specific procedures were performed
- Results of study parameters, as required by the protocol
- IP accountability records
- Documentation of AEs and other safety parameters (if applicable)
- Records regarding medical histories and the use of concomitant therapies prior to and during the study
- Date of study completion and reason for early discontinuation, if applicable

It is required that the author of an entry in the source documents be identifiable. Direct access to source documentation (medical records) must be allowed for the purpose of verifying that the data recorded on the CRF are consistent with the original source data.


Status: Effective 

Effective Date: 08-Mar-2019

Only designated individuals at the site will complete the CRFs. The CRFs must be completed at regular intervals following the clinical study visit schedule. It is expected that all data reported have corresponding entries in the source documents. The Principal Investigator is responsible for reviewing and certifying that the CRFs are accurate and complete. The only subject identifiers recorded on the CRFs will be subject number, and subject demographic information.

#### 13.3 Data Review and Clarifications

A review of CRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. After the CRFs have been completed, additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's CRF.

## 13.4 Sponsor and Monitoring Responsibilities

The Study Sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals according to the study monitoring plan. The clinical investigation will be monitored to ensure that the rights and well-being of the subjects are protected, the reported data are accurate, complete, and verifiable from the source documents, and the study is conducted in compliance with the current approved protocol (and amendments[s], if applicable), with current GCP, and with applicable regulatory requirements.

The site may not screen subjects or perform the informed consent process on any subject until it receives a notification from an appropriate Study Sponsor representative that the site may commence conducting study activities. Monitoring will be conducted periodically while the clinical study is ongoing. Monitoring methods may include site visits, telephone, written and fax correspondence. Close-out visits will take place after the last visit of the last subject at the site.

A Coordinating Investigator may be identified by the Study Sponsor to review and endorse the final study report. In cases where a Coordinating Investigator is engaged, the Study Sponsor will select the Coordinating Investigator based upon their experience, qualifications, active study participation, and their willingness and availability to take on this role.

# 13.5 Regulatory Documentation and Records Retention

The Investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the Study Sponsor and the Investigator's files will be reviewed as part of the ongoing study monitoring. Financial information is to be kept separately.


Status: Effective 

Effective Date: 08-Mar-2019

Additionally, the Investigator must keep study records and source documents consistent with the terms of the clinical study agreement with the Study Sponsor. If the Investigator retires, relocates, or for any other reason withdraws from responsibility of keeping the study records, then the Study Sponsor must be notified and suitable arrangements made for retention of study records and source documents needed to comply with national and international regulations.

## 13.6 Quality Assurance and Quality Control

The Study Sponsor will secure agreement from all involved parties to ensure direct access to all study related sites, source data and documents, and reports for the purpose of monitoring and auditing by the Study Sponsor, and inspection by domestic and foreign regulatory authorities. Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. Agreements made by the Study Sponsor with the Investigator/Institution and any other parties involved in the clinical study will be provided in writing as part of the protocol or as a separate agreement.

#### 14 ETHICS

This clinical study must be conducted in accordance with the ethical principles contained within:

- The Declaration of Helsinki, and in compliance with the ICH E6 GCP Consolidated Guideline, ISO 14155:2011, and the applicable US FDA 21 CFR Regulations.
- SOPs of the Study Sponsor and contract research organizations participating in the conduct of the clinical study and all other applicable regulations.
- Notifications and timelines for reporting protocol deviations should be based upon applicable Ethics Committee requirements

The Investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience. The Investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. Deviations from this protocol, regulatory requirements and/or GCP must be recorded and reported to the Sponsor prior to database lock. If needed, corrective and preventive action should be identified, implemented, and documented within the study records. Use of waivers to deviate from the clinical protocol is prohibited.

Before clinical study initiation, this protocol, the informed consent form, any other written information given to subjects, and any advertisements planned for subject recruitment must

Alcon - Business Use Only Effective Date: 08-Mar-2019


Status: Effective 

be approved by an IRB/IEC. The Investigator must provide documentation of the IRB/IEC approval to the Study Sponsor. The approval must be dated and must identify the applicable protocol, amendments (if any), informed consent form, assent form (if any), all applicable recruiting materials, written information for subject, and subject compensation programs. The IRB/IEC must be provided with a copy of the IB, Package Insert, any periodic safety updates, and all other information as required by local regulation and/or the IRB/IEC. At the end of the study, the Investigator must notify the IRB/IEC about the study's completion. The IRB/IEC also must be notified if the study is terminated prematurely. Finally, the Investigator must report to the IRB/IEC on the progress of the study at intervals stipulated by the IRB/IEC.

Voluntary informed consent must be obtained in writing from every subject and the process shall be documented before any procedure specific to the clinical investigation is applied to the subject. The Investigator must have a defined process for obtaining consent. Specifically, the Investigator, or their delegate, must explain the clinical study to each potential subject and the subject must indicate voluntary consent by signing and dating the approved informed consent form. The subject must be provided an opportunity to ask questions of the Investigator, and if required by local regulation, other qualified personnel. The Investigator must provide the subject with a copy of the consent form written in a language the subject understands. The consent document must meet all applicable local laws and provide subjects with information regarding the purpose, procedures, requirements, and restrictions of the study, along with any known risks and potential benefits associated with the IP and the study, the available compensation, and the established provisions for maintaining confidentiality of personal, protected health information. Subjects will be told about the voluntary nature of participation in the study and must be provided with contact information for the appropriate individuals should questions or concerns arise during the study. The subject also must be told that their records may be accessed by appropriate authorities and Sponsor-designated personnel. The Investigator must keep the original, signed copy of the consent (file in subject's medical records) and must provide a duplicate copy to each subject according to local regulations.

The Study Sponsor assures that the key design elements of this protocol will be registered on www.clinicaltrials.gov as required by current regulations and, if applicable, other public databases as required by local country regulations. In addition, results of this study will be made publicly available on www.clinicaltrials.gov regardless of outcome as required by current regulations and, if applicable, in other public databases as required by local country regulations.


Status: Effective 

Effective Date: 08-Mar-2019

# 15 REFERENCES

## 15.1 References applicable for all clinical studies

 ISO 11980:2012 Ophthalmic optics - Contact lenses and contact lens care products -Guidance for clinical investigations

 ISO 14155:2011 Clinical investigation of medical devices for human subjects - Good clinical practice

# 15.1.1 US references applicable for clinical studies

- 21 CFR Part 11 Electronic Records; Electronic Signatures
- 21 CFR Part 50 Protection of Human Subjects
- 21 CFR Part 56 Institutional Review Boards
- 21 CFR Part 812 Investigational Device Exemptions
- 21 CFR Part 54 Financial Disclosure by Clinical Investigators
- The California Bill of Rights

## 15.2 References for this clinical study

Morgan PB, Woods CA, Tranoudis IG, Efron N, Jones L, Aighamdi W, et al. International contact lens prescribing in 2018. Contact Lens Spectrum. 2019 (Jan);34:26-32.


Effective Date: 08-Mar-2019

Status: Effective

Document: TDOC-0056081